CLINICAL TRIAL: NCT07313462
Title: Escalation vs. Induction Therapy Strategy in Patients With Early-Onset MS After Age 50
Acronym: 50-CENT
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9535
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple Sclerosis (MS); Escalation Therapy; Induction Therapy
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The objective of this study is to evaluate the risk of inflammatory disease activity by retrospectively comparing two therapeutic strategies (escalation group and induction group). The investigators also aim to identify factors associated with inflammatory relapse and treatment-related complications.

ELIGIBILITY:
Inclusion Criteria:

* Patients with RRMS onset after age 50
* Patients who started their first disease-modifying therapy within 2 years of the first symptoms
* Patients Treated with moderately effective disease-modifying antirheumatic drugs (DMARDs) (teriflunomide, dimethyl fumarate or diroximel fumarate, glatiramer acetate, interferon beta, peginterferon)
* Patient treated with highly effective DMARDs (fingolimod, ponesimod, natalizumab, rituximab, ocrelizumab, ofatumumab, cladribine)

Exclusion Criteria:

- Patients with early progressive MS

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with RRMS onset after age 50
Sampling Method: Non-Probability Sample
Enrollment: 830 (Estimated)
Dates: Start 2025-02-07 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Time to First Clinical Inflammatory Relapse | Up to 12 months
  Compare the time to first clinical inflammatory relapse between two groups of patients who developed relapsing-remitting MS (RRMS) after age 50:
  * Group 1 = therapeutic escalation strategy: starting with a moderately effective treatment (teriflunomide, dimethyl fumarate or diroximel fumarate, glatiramer acetate, interferon beta, peginterferon)
  * Group 2 = induction strategy: starting with a highly effective treatment (fingolimod, ponesimod, natalizumab, rituximab, ocrelizumab, ofatumumab, cladribine)

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Investigation Clinique - CHU de Strasbourg - France, Strasbourg, France